CLINICAL TRIAL: NCT04378777
Title: A Prospective Cohort Study to Assess Longitudinal Immune Responses in Hospitalized Patients With COVID-19 (DAIT-COVID-19-002)
Brief Title: Immunophenotyping Assessment in a COVID-19 Cohort
Acronym: IMPACC
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Benaroya Research Institute (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT-COVID-19-002; NIAID CRMS ID#: 38733 (Other: DAIT NIAID)
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus Disease 2019 (COVID-19); SARS-CoV-2
Keywords: observational cohort surveillance study; immunologic assessments
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * nasal secretion samples
  * whole blood
  * sputum secretions by endotracheal aspiration (for intubated patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surveillance cohort: Cohort descriptive data will include demographic variables (e.g. age, sex, race, ethnicity), clinical information on enrollment and key aspects of medical history (e.g. concomitant medications, for example). Patients will be longitudinally followed, up to 12 months.
  Interventions: Procedure: Biological sample collection; Procedure: Data Collection: Clinical Care Assessments

INTERVENTIONS:
Procedure: Biological sample collection — During patient hospitalization: Nasal secretion samples by nasal swabs (for non-intubated patients), whole blood (blood draw/phlebotomy) and sputum secretions by endotracheal aspiration (for intubated patients) will be obtained to proceed with immunologic analysis of samples. DNA will be collected from whole blood at enrollment for genetic analysis (e.g., genome-wide association study [GWAS]). After hospital discharge: Collection of biologic samples (involving nasal swabs and blood draw/phlebotomy) will occur up to 12 months.
Procedure: Data Collection: Clinical Care Assessments — Baseline data and assessments obtained as part of ongoing clinical care will be collected throughout hospitalization for COVID-19. After hospital discharge, clinical status and activity assessments will occur up to 12 months.
  Other Names: Baseline data, clinical care assessments

SUMMARY:
This surveillance study will collect detailed clinical, laboratory, and radiographic data in coordination with biologic sampling of blood and respiratory secretions and viral shedding in nasal secretions in order to identify immunophenotypic and genomic features of COVID-19 -related susceptibility and/or progression. The aim: for the results obtained from this study to assist in generating hypotheses for effective host-directed therapeutic interventions, to help to prioritize proposals for such interventions, and/or optimize timing for administration of host-response directed therapeutics.

DETAILED DESCRIPTION:
This is a prospective observational cohort surveillance study of up to 2,000 adult participants hospitalized with known or presumptive COVID-19. Detailed information will be collected regarding patient history and onset of illness upon enrollment. Participants will undergo longitudinal assessments of clinical status and pertinent clinical data (including clinical laboratory values, radiographic findings, medication use, oxygen and ventilatory support requirements, complications, etc.) will be recorded. In parallel, the study will conduct serial biologic sampling for detailed immunophenotyping to provide a comprehensive picture of immune changes that occur throughout the course of infection. The biologic samples to be collected for this observational study include blood, nasal swabs, and endotracheal aspirates.

Participants will be followed in hospital through Day 28, unless discharged earlier. If a participant requires an escalation to Intensive Care Unit (ICU)-level care, either within or outside of a dedicated ICU, additional samples will be collected within 24 and 96 hours of care escalation. Convalescent questionnaires and biologic samples will be collected at 3-month intervals up to Month 12 after infection symptom onset, if available. In addition, if a participant is discharged from the hospital prior to Day 28, attempts will be made to collect additional scheduled assessments through Day 28 on an outpatient basis, if feasible.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

* Participant and/or surrogate understands the data to be collected and the study procedures and is willing to participate in the surveillance cohort as described in the study information sheet;
* ≥ 18 years of age at the time of hospitalization; and
* Admitted to a hospital with presumptive or documented coronavirus disease 2019 (COVID-19), with confirmation of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) infection by Polymerase Chain Reaction (PCR).

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

* Underlying medical problems which, in the opinion of the investigator may be associated with mortality unrelated to COVID-19 within 48 hours of hospitalization, or a decision by the patient or surrogate prior to hospitalization to limit care to comfort measures; or
* Medical problems or conditions such as pregnancy which might impact interpretation of the immunologic data obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult participants hospitalized with known or presumptive coronavirus disease 2019 (COVID-19), a human disease caused by Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) infection.
Sampling Method: Non-Probability Sample
Enrollment: 1227 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Mortality Rate Among COVID-19 Patients | Day 1 to Day 28
  The incidence of mortality in the first 28 days.
Proportion of Patients with COVID-19 who Require Intensive Care Unit (ICU)-Level Care, Mechanical Ventilatory Support (MV), and/or Extracorporeal Membrane Oxygenation (ECMO) Over Time to Day 28 | Day 1 to Day 28
  As a measure of disease acuity and severity.
Proportion of Patients with COVID-19 who Develop Shock, Secondary Organ Failure, or Secondary Infection Over Time to Day 28 | Day 1 to Day 28
  As a measure of disease acuity and severity.
Mechanistic: Longitudinal Assessment of Viral Load by Semi-Quantitative Polymerase Chain Reaction (PCR) Over Time to Day 28 | Day 1 to Day 28
  Ribonucleic acid (RNA) from the nasal swab will be used to assess SARS-CoV-2 viral load.
Mechanistic: Antibody Isotype/Subclass Classification and Functionality Over Time through Day 28 and at follow-up through month 12 | Up to 12 Months
  Focus on the immune response to SARS-CoV-2, seroconversion and immunoglobulin and transitions. Antibody isotypes present in a patient specimen(s) provide information about the timing of initial exposure and may provide insight on the progression of the disease and prognosis.
Mechanistic: Longitudinal Assessment of Inflammatory Mediators as Collected Over Time to Day 28 | Day 1 to Day 28
  Collected as part of clinical care.
Mechanistic: Longitudinal Assessment of Markers of Myocardial Injury Over Time to Day 28 | Day 1 to Day 28
  Collected as part of clinical care.

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation in Patients with COVID-19 Over Time to Day 28 | Day 1 to Day 28
  A measure of disease morbidity.
Proportion of Patients with COVID-19 with Requirement for New (Or Increased from Baseline if on Home Oxygen) Supplemental Oxygen Over Time to Day 28 | Day 1 to Day 28
  A measure of disease morbidity.
Requirement for Extracorporeal Membrane Oxygenation (ECMO) in COVID-19 Patients with COVID-19 Over Time to Day 28 | Day 1 to Day 28
  A measure of disease morbidity.
Mechanistic: Immune Cell Frequencies and Activation Status (CyTOF) in Blood and Endotracheal Aspirate over time Through Day 28 and In blood at Select Study Visits Through Month 12 | Up to 12 Months
  Method of immune profiling and quantitating the response to COVID-19 over time.
Mechanistic: Gene Expression (Transcriptomics) in Blood | Up to 12 Months
  To identify and quantitate differences in immune response associated with disease outcome.
Mechanistic: Gene Expression (Transcriptomics) in Respiratory Epithelium | Up to 12 Months
  To identify and quantitate differences in immune response associated with disease outcome.
Mechanistic: Gene Expression (Transcriptomics) in Plasma Protein | Up to 12 Months
  To identify and quantitate differences in immune response associated with disease outcome.
Mechanistic: Gene expression (Transcriptomics) in Metabolic Profiling | Up to 12 Months
  To identify and quantitate differences in immune response associated with disease outcome.
Mechanistic: Circulating Immune Mediators Assessed by OLINK Methodology | Up to 12 Months
  Circulating immune biomarkers will be explored by use of the OLINK® (name of brand), a multiplex protein biomarker discovery panel.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, M.D., Study Chair — Emory University
Locations (17):
- United States (17):
  - University of Arizona (UA) College of Medicine - Tucson: UA Health Sciences Asthma and Airway Disease Research Center, Tucson, Arizona
  - University of California, Los Angeles: Department of Medicine, Los Angeles, California
  - University of California San Francisco School of Medicine, San Francisco, California
  - Stanford Medicine: Sean N. Parker Center for Allergy & Asthma Research, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida Health Gainesville, Gainesville, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of South Florida Health Tampa, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Oklahoma ,Oklahoma Health Sciences Center: Pulmonary/Critical Care, Department of Medicine, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Texas at Austin: UT Health Austin, Austin, Texas
  - Baylor College of Medicine: Department of Medicine, Houston, Texas

REFERENCES:
- [Derived] Gabernet G, Maciuch J, Gygi JP, Moore JF, Hoch A, Syphurs C, Chu T, Doni Jayavelu N, Corry DB, Kheradmand F, Baden LR, Sekaly RP, McComsey GA, Haddad EK, Cairns CB, Rouphael N, Fernandez-Sesma A, Simon V, Metcalf JP, Agudelo Higuita NI, Hough CL, Messer WB, Davis MM, Nadeau KC, Pulendran B, Kraft M, Bime C, Reed EF, Schaenman J, Erle DJ, Calfee CS, Atkinson MA, Brakenridge SC, Melamed E, Shaw AC, Hafler DA, Augustine AD, Becker PM, Ozonoff A, Bosinger SE, Eckalbar W, Maecker HT, Kim-Schulze S, Steen H, Krammer F, Westendorf K; IMPACC Network; Peters B, Fourati S, Altman MC, Levy O, Smolen KK, Montgomery RR, Diray-Arce J, Kleinstein SH, Guan L, Ehrlich LI. A multiomics recovery factor predicts long COVID in the IMPACC study. J Clin Invest. 2025 Sep 9;135(21):e193698. doi: 10.1172/JCI193698. eCollection 2025 Nov 3. PMID 40924481
- [Derived] Gygi JP, Maguire C, Patel RK, Shinde P, Konstorum A, Shannon CP, Xu L, Hoch A, Jayavelu ND, Haddad EK; IMPACC Network; Reed EF, Kraft M, McComsey GA, Metcalf JP, Ozonoff A, Esserman D, Cairns CB, Rouphael N, Bosinger SE, Kim-Schulze S, Krammer F, Rosen LB, van Bakel H, Wilson M, Eckalbar WL, Maecker HT, Langelier CR, Steen H, Altman MC, Montgomery RR, Levy O, Melamed E, Pulendran B, Diray-Arce J, Smolen KK, Fragiadakis GK, Becker PM, Sekaly RP, Ehrlich LI, Fourati S, Peters B, Kleinstein SH, Guan L. Integrated longitudinal multiomics study identifies immune programs associated with acute COVID-19 severity and mortality. J Clin Invest. 2024 May 1;134(9):e176640. doi: 10.1172/JCI176640. PMID 38690733
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait